CLINICAL TRIAL: NCT02629679
Title: Prospective Analysis of the Factors Associated With Substance Use and Misuse in Adolescents
Brief Title: Sports, Education and Consumption of Substances in Adolescents
Acronym: SESA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Split (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Damir Sekulic, Professor Damir Sekulic, University of Split
Other Study IDs: 01111705/2015
Record Dates: First submitted 2015-12-02; First posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Cigarette Smoking; Alcohol Drinking
MeSH Terms: conditions — Cigarette Smoking; Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Males nonathletes: Boys non-involved in organized sport and exercising
  Interventions: Behavioral: Regular scholastic system
- Females nonathletes: Girls non-involved in organized sport and exercising
  Interventions: Behavioral: Regular scholastic system
- Males athletes: Athletic boys (involved in sports)
  Interventions: Behavioral: Regular scholastic system and organized sports
- Females athletes: Athletic girls (involved in sports)
  Interventions: Behavioral: Regular scholastic system and organized sports

INTERVENTIONS:
Behavioral: Regular scholastic system and organized sports — This group will consist of children involved in regular school system who at the same time participate in organized sport in sport-clubs
  Groups: Females athletes; Males athletes
Behavioral: Regular scholastic system — The group will consist of children who are regularly in school, but not being involved in organized sport activities
  Groups: Females nonathletes; Males nonathletes

SUMMARY:
Adolescent substance abuse (SA), which includes the consumption of alcohol, cigarette smoking, the consumption of drugs and other behaviors, is a significant public-health issue in the world today. Recent data showed that prevalence of SA among adolescents in Croatia and surrounding countries (i.e. former Yugoslav republics) is alarming and needs serious intervention. It is hypothesized that participation in physical-exercise-and-sport (PE&S) will reduce the tendency of young people to abuse substances. However, the literature to date has not consistently validated the perception PE&S factors are factors which could buffer SA among children and adolescents. One of the probable reasons for evident inconsistencies on findings about relationship between PE&S and SA is a cross-sectional nature of studies done so far. Therefore, the main rationale (i.e. problem) of this study is lack of current knowledge about influence of the PE&S on SA among adolescents. The main objective of this study is to prospectively investigate the influence of PE&S on SA among adolescents aged 17 to 18 years old. Aims of the project are: (1) to define prevalence and trends of SA among adolescents aged 17 to 18 years old; (2) to define prevalence and trends of PE&S participation; (3) to establish interrelationships which exist between socio-demographic, psychological, educational-factors, and PE&S (predictors); (4) to identify multivariate and univariate associations between: socio-demographic and SA, psychological factors and SA, PE&S and SA, educational - scholastic factors and SA.Expected results of the project are: (1) definition of the prevalence of SA among adolescents; (2) definition of the adolescents' participation in PE&S; (3) identification and interpretation relationships which exist between and within studied predictors of SA (educational factors, socio-demographic factors, PE&S, psychological factors); (4) identification of the influence of studied predictors on SA.

ELIGIBILITY:
Inclusion Criteria:

* Children involved in regular scholastic system

Exclusion Criteria:

* No

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample will comprise approximately 1,000 participants (50% males). At the beginning of the study, the participants will be attending the 3rd year (grade) of high school, and therefore practically all subjects will be 17 years of age at the moment the study starts (+/- 6 months). Participants will be randomly selected from 10 to 15 high schools which offer a 4-year high school education. Because of the prospective study design and consequent need to repeatedly test the same participants, only those schools where the investigators already have personal and professional contacts with the school authorities will be used as possible test environments.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Exact number of participants who smoke cigarettes as assessed by QSU questionnaire | 2 years
  QSU - Questionnaire of Substance Use is validated questionnaire where participants are asked on their consumption of substances, including cigarette smoking
Exact number of participants involved in harmful alcohol drinking as assessed by AUDIT questionnaire | 2 years
  AUDIT - Alcohol Use Disorders Identification Test is a common and valid questionnaire where subjects are tested on alcohol drinking habits

SECONDARY OUTCOMES:
Exact number of participants who failed educationally as assessed by grade-point average | 2 years
  Grade-point-average is one of the scholastic-achievement variables.
Exact number of participants who failed educationally as assessed by behavioral grade | 2 years
  Behavioral-grade is one of the scholastic-achievement variables.

REFERENCES:
- [Background] Zenic N, Ostojic L, Sisic N, Pojskic H, Peric M, Uljevic O, Sekulic D. Examination of the community-specific prevalence of and factors associated with substance use and misuse among Rural and Urban adolescents: a cross-sectional analysis in Bosnia and Herzegovina. BMJ Open. 2015 Nov 6;5(11):e009446. doi: 10.1136/bmjopen-2015-009446. PMID 26546145
- [Background] Zenic N, Terzic A, Rodek J, Spasic M, Sekulic D. Gender-Specific Analyses of the Prevalence and Factors Associated with Substance Use and Misuse among Bosniak Adolescents. Int J Environ Res Public Health. 2015 Jun 10;12(6):6626-40. doi: 10.3390/ijerph120606626. PMID 26068091
- [Background] Idrizovic K, Zenic N, Tahirajl E, Rausavljevic N, Sekulic D. CIGARETTE SMOKING AMONG 17-18 YEAR OLD ADOLESCENTS - PREVALENCE AND ASSOCIATION WITH SOCIODEMOGRAPHIC, FAMILIAL, SPORT, AND SCHOLASTIC. FACTORS. Med Pr. 2015;66(2):153-63. doi: 10.13075/mp.5893.00104. PMID 26294308
- [Background] Sekulic D, Ostojic M, Ostojic Z, Hajdarevic B, Ostojic L. Substance abuse prevalence and its relation to scholastic achievement and sport factors: an analysis among adolescents of the Herzegovina-Neretva Canton in Bosnia and Herzegovina. BMC Public Health. 2012 Apr 5;12:274. doi: 10.1186/1471-2458-12-274. PMID 22480230
- [Background] Modric T, Zenic N, Sekulic D. Substance use and misuse among 17- to 18-year-old Croatian adolescents: correlation with scholastic variables and sport factors. Subst Use Misuse. 2011;46(10):1328-34. doi: 10.3109/10826084.2011.579677. Epub 2011 May 25. PMID 21612340